CLINICAL TRIAL: NCT06952764
Title: Epilepsy Cycles Longitudinal Monitoring to Inform Personalized Seizure-risk Estimation, A Double-blinded Study of Seizure Forecasting and Randomized Information Withdrawal in Adults With Epilepsy.
Brief Title: Epilepsy Cycles Longitudinal Monitoring to Inform Personalized Seizure-risk Estimation (ECLIPSE)
Acronym: ECLIPSE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2025 - SWEZ01
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy (Treatment Refractory)
Keywords: Seizure forecasting
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Three sequential phases:
  1. Covert phase: double-blinded (participant, investigator)
  2. Overt phase: open-label
  3. Withdrawal phase: double-blinded (participant, investigator), randomized, controlled, cross-over withdrawal of seizure forecast
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IEEG-forecast (Experimental): Potentially informative seizure forecast.
  Interventions: Other: Seizure risk forecast
- Control-forecast (Active Comparator): Uninformative control seizure forecast.
  Interventions: Other: Control seizure risk forecast

INTERVENTIONS:
Other: Seizure risk forecast — Participants are provided with daily risk estimates about upcoming seizure likelihood.
  Arms: IEEG-forecast
Other: Control seizure risk forecast — Participant receive uninformative control forecast
  Arms: Control-forecast

SUMMARY:
The occurrence of seizures in epilepsy is not entirely random. Temporal patterns that organize the occurrence of seizures over weeks and months were previously unraveled using intracranial EEG System (IEEG) that monitors epileptic brain activity chronically. Seizures typically recur with patient-specific periodicity and are preceded by increases of epileptic brain activity over days. Here, the investigators developed new methods to forecast seizure likelihoods at a 24-h horizon. In this trial, participants will be provided with daily estimates about their upcoming risk of seizures. As a primary outcome, the performance of forecasts will be evaluated against the occurrence of electrographic seizures. As secondary outcome, the forecast's potential benefit for users in conveying actionable information in real-life will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adult with diagnosed pharmacoresistant epilepsy and at least one self-reported seizure in the last 12 months.
* Patients previously implanted with the RNS System, on stable detection settings enabling reliable detection of electrographic seizures.
* Patients willing and able to keep a diary, issue self-forecasts, and follow instructions.
* Home equipped with an internet connection.
* Informed Consent signed by the subject

Exclusion Criteria:

* Insufficient number of electrographic seizures or insufficient forecasting performance in the training phase.
* Women pregnant at the time of recruitment (later pregnancy not a contra-indication)
* Subjects with a history of psychogenic non-epileptic seizures
* Clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.)
* Vulnerable subjects, including severe cognitive impairment precluding informed consent
* Drug or alcohol addiction
* Subjects who are unable (i.e., mentally or physically impaired patients) or do not have the necessary assistance, to properly operate the device system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Forecast performance | At least on the first 10 seizures since enrollment. Expected within 6-12 months from enrollment.
  Performance of double-blinded (covert phase) IEEG-forecasts. Performance is quantified as the area-under-the sensitivity vs. time in warning curve (AUC) and double-tested statistically in a pairwise manner against shuffled chance-forecasts and participant's self-forecasts.

SECONDARY OUTCOMES:
Maintenance of forecast performance | At least 8 seizures during the overt phase, expected to last 6-12 months
  For the cohort that progresses to the overt phase, The AUC obtained during the overt phase will be compared to their historical AUC during the covert phase and tested for a pairwise difference.
Informativity | Throughout the open-label (6-12 months) and withdrawal phase (3-6 months)
  Participant-reported estimates of how informative a forecast is on a visual-analogue scale, scored from 0 to 10.
QOLIE-31 | Upon completion of the study after 18-30 months.
  Quality Of Life In Epilepsy questionnaires with 31 items (QOLIE-31) completed at the transition from one study phase to the next. The quantification is on a scale from 0 to 100 and pairwise comparison between covert, overt and withdrawal phase.
Actionability | End of open-label phase after 12-24 months.
  List of concrete strategies enabled by the forecasts

OTHER OUTCOMES:
Seizure rate | Upon completion of each phase, after 6-12, 12-24 and 18-30 months.
  Participant's seizure rate in each phase of the trial expressed as the probability of a seizure per day.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime O Baud, MD, PhD, Study Chair — Department of Neurology, Inselspital Bern
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data can be shared by the investigators upon study completion based on a reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be shared 2-4 years after study start and up to a duration of 10 years.
Access Criteria: Researcher will be able to access the data.